CLINICAL TRIAL: NCT00494949
Title: A Clinical Safety (Phase Ib/II) Increasing Dose Study of MP4 (Hemospan) in Orthopedic Surgery Patients
Brief Title: Increasing Dose Safety Study of Hemospan in Orthopedic Surgery Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3002
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Hypotension; Hypoxia
Keywords: Anesthesia, spinal; Blood substitutes; Oxygen therapeutics; Orthopedic surgery; Plasma expanders; Vasoconstriction; Hemospan
MeSH Terms: conditions — Hypotension; Hypoxia | interventions — maleimide-polyethylene glycol-modified hemoglobin, MP4; Ringer's Lactate; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemospan (MP4OX) (Experimental): 4.3 g/dL MalPEG-Hb solution
  Interventions: Drug: Hemospan (MP4OX)
- Control (Active Comparator): Ringer's lactate
  Interventions: Drug: Ringer's lactate

INTERVENTIONS:
Drug: Hemospan (MP4OX) — 200, 400, 600, 750, or 1000 mL of Hemospan (MP4OX)
  Other Names: MP4OX solution; 4.3 g/dL MalPEG-Hb; PEGylated Hb
  Arms: Hemospan (MP4OX)
Drug: Ringer's lactate — 200, 400, 600, 750, or 1000 mL of Ringer's lactate solution
  Other Names: Lactated Ringers; Ringers solution; Hartmann's solution
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the safety and possible effectiveness of Hemospan solution in patients undergoing elective orthopedic surgery who receive spinal anesthesia.

DETAILED DESCRIPTION:
Allogeneic (donor) blood transfusions are often required during and/or after orthopedic hip surgery to maintain adequate hemoglobin concentration, prevent tissue ischemia, treat hypotension, and compensate for fluid shifts. For example, during hospitalization for hip replacement, patients may receive up to two to three units of blood. This amount varies depending on the technical difficulty of the surgery, the patient's hemoglobin concentration prior to surgery, and the patient's clinical status.

The limited availability, logistic constraints and documented risks associated with allogeneic blood transfusions have prompted the search for alternative therapies. Autologous (self-donated) red blood cell pre-donation can be used in many cases but age, anemia and co-morbidities often preclude the use of this treatment. Cell saving and re-infusion also prevents blood transfusion, but this practice also has potential problems and limited applicability.

Over the past 75 years various "blood substitutes" have been developed for potential clinical use. To date all have shown significant toxicity in preclinical or clinical studies and regulatory approval of these synthetic or hemoglobin-based products has been impeded by safety concerns.

Hemospan is a novel polyethylene-modified hemoglobin solution specifically developed to perfuse and oxygenate tissue at risk for ischemia and hypoxia. As a result of the molecular size and oxygen dissociation characteristics, Hemospan selectively off-loads oxygen in tissues predisposed to low oxygen tension. In preclinical studies Hemospan has been found to be free of significant toxicity in a variety of animal species in doses exceeding those that will be used in this study.

In the Phase I safety study in normal volunteers, Hemospan was well tolerated in doses up to 100 mg/kg (approximately 200 mL of a 4g/dL Hemospan solution).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or postmenopausal female(last menses at least 12 months prior and laboratory assessment verifying appropriate FSH and LH levels [laboratory assessments not necessary if last menses at least 12 months prior]), American Society of Anesthesiologists classification system (ASA) class I or II patients over the age of 18 scheduled for orthopedic surgery with spinal anesthesia
* Patients have to be in good health (other than the orthopedic indication for surgery) as determined by medical history, physical examination, clinical laboratory studies and ECG, all within four weeks prior to drug administration
* At screening (within four weeks prior to drug administration) the iohexol clearance, urinalysis and hematology (hemoglobin, hematocrit, RBC, WBC, platelets, reticulocytes percentage), PT, PTT had to be within the laboratory normal limits, If a clinical laboratory value (Na, K, albumin, serum creatinine, urea, bilirubin, AST, ALT, ALP, GGT, LDH, conjugated bilirubin, lipase, amylase, total protein, C1, Ca, CK, CK-MB, troponin, cholesterol, glucose, β-2 microglobulin, NAG, osmolarity) is outside the normal range the laboratory test can be repeated. A patient with two consecutive abnormal values is not allowed to participate in the study unless the PI determines the change is not clinically significant. A notation of "Not clinically significant (NCS)" is noted on the laboratory record in that case.
* Patients have to sign an informed consent form for the study, which is reviewed and approved by the IECs of the Karolinska Hospital or the Stockholm Söder Hospital

Exclusion Criteria:

* Any acute or chronic condition which limits the patient's ability to complete the study or jeopardizes the safety of the patient
* Patients with a history, or clinical manifestation of significant metabolic disorders, cardiovascular disorders (including arrhythmia, tachycardia, hypertension, angina pectoris, chronic heart failure) or psychiatric disorders
* Patients with a history of chronic hepatic or renal disease
* Pregnancy
* Patients who have received any other investigational drugs within 30 days prior to administration of the study drug
* Patients who test positive to human immunodeficiency virus (HIV), hepatitis B or hepatitis C screens or have any other chronic infection
* Professional or ancillary personnel involved with the study
* Presence of a hemoglobinopathy
* Known allergy to iodine-containing intravenous contrast material or seafood
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-04; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 21 days

SECONDARY OUTCOMES:
Changes from baseline in pulse oximetry | 4 days
Change in Arterial blood gas and blood lactate levels from baseline | 4 days
Duration of supplemental inspired oxygen [FIO2] | 4 days
Number and duration of intra-operative hypotensive episodes (SBP<90 mmHg or a DBP <50 mmHg) | 4 days
Incidence of pharmacologic intervention for hypotension | 4 days
Volume blood products administered | 4 days
Change from baseline in vital signs | 4 days
Changes in serum chemistry and hematology from baseline | 4 days
Volume of IV fluids given | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Christina I. Olofsson, MD, PhD, Principal Investigator — Karolinska University Hospital, Stockholm
Locations (2):
- Sweden (2):
  - Department of Orthopedics, Karolinska Hospital, Stockholm
  - Department of Orthopedics, Stockholm Söder Hospital, Stockholm

REFERENCES:
- [Background] Bjorkholm M, Fagrell B, Przybelski R, Winslow N, Young M, Winslow RM. A phase I single blind clinical trial of a new oxygen transport agent (MP4), human hemoglobin modified with maleimide-activated polyethylene glycol. Haematologica. 2005 Apr;90(4):505-15. PMID 15820947
- [Background] Winslow RM. Red cell substitutes. Semin Hematol. 2007 Jan;44(1):51-9. doi: 10.1053/j.seminhematol.2006.09.013. PMID 17198847
- [Result] Olofsson C, Ahl T, Johansson T, Larsson S, Nellgard P, Ponzer S, Fagrell B, Przybelski R, Keipert P, Winslow N, Winslow RM. A multicenter clinical study of the safety and activity of maleimide-polyethylene glycol-modified Hemoglobin (Hemospan) in patients undergoing major orthopedic surgery. Anesthesiology. 2006 Dec;105(6):1153-63. doi: 10.1097/00000542-200612000-00015. PMID 17122578
- See also: Click here for more information about Sangart — http://www.sangart.com